CLINICAL TRIAL: NCT05400460
Title: Outcomes Under Three Different Procedures for Anterior Cruciate Ligament Reconstruction, a Prospective Randomized Cohort Study
Brief Title: Prognosis Study of Different Anterior Cruciate Ligament Surgery Methods
Acronym: ACLRSurgRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu Jiakuo (Other)
Responsible Party: Sponsor-Investigator, Yu Jiakuo, Clinical Professor, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACLSurgRCT-20160601
Record Dates: First submitted 2022-05-01; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior cruciate ligament (ACL); Signal of noise (SNQ); Graft bending angle (GBA); Central axial single-bundle; Anatomical single-bundle; Double bundle
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Prospective randomized cohort of patients with anterior cruciate ligament rupture assigned to three procedures and followed up two years after surgery.In this trial, patients diagnosed with anterior cruciate ligament rupture in the outpatient clinic were randomly assigned to the following three procedures: central axial single-bundle reconstruction (CASBR), anatomical single-bundle reconstruction (ASBR), and double-bundle reconstruction (DBR).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASBR group (Other): Anterior cruciate ligament reconstruction using STG, absorbable interface nails and ASBR procedures.
  Interventions: Procedure: Anatomical single-bundle reconstruction（ASBR method）; Other: rehabilitation training protocol; Other: Educate patients on return to sports and the importance of quadriceps strength
- CASBR group (Other): Anterior cruciate ligament reconstruction using STG, absorbable interface nails and CASBR procedures.
  Interventions: Procedure: Central axial single-bundle reconstruction（CASBR group）; Other: rehabilitation training protocol; Other: Educate patients on return to sports and the importance of quadriceps strength
- DB group (Other): Anterior cruciate ligament reconstruction using STG, absorbable interface nails and DBR procedures.
  Interventions: Procedure: Double-bundle reconstruction （DBR method）; Other: rehabilitation training protocol; Other: Educate patients on return to sports and the importance of quadriceps strength

INTERVENTIONS:
Procedure: Anatomical single-bundle reconstruction（ASBR method） — 406 people were enrolled in the outpatient clinic, after screening for inclusion and exclusion. Of the remaining 243 patients who participated in this RCT, 81 were randomly assigned to the ASBR group to receive anatomic single-bundle reconstruction.We used hamstring as an autograft in the operation, and we chose the anatomical footprint of the anterior cruciate ligament for the positioning of the bone tunnel.Arthroscopic ASB ACL reconstruction was conducted with AMP technique.
  Other Names: ASB
  Arms: ASBR group
Procedure: Double-bundle reconstruction （DBR method） — 406 people were enrolled in the outpatient clinic, after screening for inclusion and exclusion. Of the remaining 243 patients who participated in this RCT, 81 were randomly assigned to the DBR group to receive double bundle reconstruction.The hamstring autograft is still used for double-bundle reconstruction. The surgical approach is to treat the native ligaments as anteromedial bundles and posterolateral bundles and restore the structure of the two bundles of ligaments in the process of a
  Other Names: DB
  Arms: DB group
Procedure: Central axial single-bundle reconstruction（CASBR group） — 406 people were enrolled in the outpatient clinic, after screening for inclusion and exclusion. Of the remaining 243 patients who participated in this RCT, 81 were randomly assigned to CASBR group.Arthroscopic ASB ACL reconstruction was conducted with transtibial technique and using Hamstring as autograft.Single-bundle reconstruction is used in CASBR reconstruction surgery.
  The footprint of the implant on the lateral femoral condyle was chosen to be the location of the AMB bone canal in DB reconstruction surgery while the footprint of the implant on the tibial plateau was chosen to be the location of the bone canal of the PLB in DB reconstruction surgery.
  Other Names: CASB
  Arms: CASBR group
Other: rehabilitation training protocol — The rehabilitation program for all patients followed a standardized Process. The first day after surgery, quadriceps sets, straight-leg raises, and prone hangs were initiated. All of the patients were allowed to walk with crutches and braces but with no weightbearing. The range of motion (ROM) progressed from 0 to 90 degrees 3 to 7 days postoperatively and reached 115 degrees within fourth week. Closed kinetic chain exercises and full weightbearing were started in the sixth week. Patients progressed to running without braces at 4 to 6 months.
Other: Educate patients on return to sports and the importance of quadriceps strength — Patients were interviewed by telephone preoperatively, 6 months postoperatively, and 1 year postoperatively to ask about Tegner scores and to encourage reasonable return to sports from 6 months postoperatively.
  Inform patients of the possibility of osteoarthritis in patients undergoing ACL reconstruction preoperatively, 6 months postoperatively, and 1 year postoperatively in telephone interviews.Tell the patient that return to sports and quadriceps strength is a must if the knee cartilage damage is to improve.

SUMMARY:
From June 1, 2016, to July 1, 2017, a total of 406 patients with ACL rupture were randomly assigned to three different ACL surgeries: anatomical single-bundle, central axial single-bundle and double-bundle. A prospective randomized cohort study was conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-45.
2. ACL rupture confirmed by both physical examination and MRI.
3. Surgery done by senior doctor.
4. Using STG as autograft.

Exclusion Criteria:

1. With bilateral acl rupture.
2. Second injury.
3. Previous surgery in extremity.
4. With OA.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 406 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2021-01-17 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging (MRI) to assess graft healing | At 2 years after surgery
  The difference in signal density between reconstructed ACL and PCL was used to measure graft ligamentation on MRI. Higher signal values represent higher inflammation and lower signal values represent better ligamentation.
Quadriceps strength | At 2 years after surgery
  Side to side quadriceps strength assessed by Biodex arthrometer test
Knee laxity （physical exam） | At 2 years after surgery
  The side to side knee joint laxity of patients after anterior cruciate ligament surgery can be divided into four grades: grade A: -1~2mm(0+), grade B: 3~5mm (1+), grade C: 6~10mm (2+) and D Grade: >10mm(3+) assessed by Lachman test of physical examination.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 2 years after surgery
  Patients will be asked to fill out the IKDC2000 score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee laxity （KT-2000 arthrometer） | At 2 years after surgery
  The knee laxity test of the forward KT-2000 measured knee laxity at pressures of 132Nt, 88Nt, 66Nt, and 44Nt, respectively, while the back-pushing KT-2000 was measured at -132NT, 88Nt, 66Nt, and -44Nt. The foward-pushing KT-2000 asessed side-to-side can be stratified into five levels are (A) < - 1 mm, (B) - 1 to 1 mm, (C) 1-3 mm, (D) 3-5 mm and (E) > 5 mm.
  The back-pushing KT-2000 is also divided into side to side differences as (A) < - 2 mm, (B) - 2 to - 0.5 mm, (C) - 0.5 to 0.5 mm, (D) 0.5-1 mm and ( E) > 1 mm.
Magnetic resonance imaging (MRI) | At 2 years after surgery
  Magnetic resonance was used to calculate the graft bending angle (GBA), which is the angle between the intra-femoral graft and the intra-articular graft. GBA is associated with graft widening and graft healing.
Magnetic resonance imaging (MRI) | At 2 years after surgery
  We used magnetic resonance 3D reconstruction to derive the area perpendicular to the bony canal and subdivide it into the proximal, mid and distal bony canal of the tibia and femur. Since CT is harmful to the human body, we used magnetic resonance imaging instead of CT to collect the last follow-up data of bone tract widening during the return visit.

SECONDARY OUTCOMES:
Gender | At baseline
  Measuring whether gender is a risk factor for anterior cruciate ligament reconstruction failure
Age | At baseline
  Measuring whether age is a risk factor for anterior cruciate ligament reconstruction failure
BMI | At baseline
  Weight and height will be combined to report BMI in kg/m^2. Measuring whether bmi is a risk factor for anterior cruciate ligament reconstruction failure
Single-Legged Hop Test | At 2 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the single hop for distance.
Single-Legged Hop Test | At 5 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the single hop for distance.
Single-Legged Hop Test | At 10 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the single hop for distance.
Triple hop test | At 2 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the triple hop for distance.
Triple hop test | At 5 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the triple hop for distance.
Triple hop test | At 10 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the triple hop for distance.
Cross hop test | At 2 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the cross hop for distance.
Cross hop test | At 5 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the cross hop for distance.
Cross hop test | At 10 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the cross hop for distance.
6-m hop test | At 2 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the 6-meter hop for time.
6-m hop test | At 5 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the 6-meter hop for time.
6-m hop test | At 10 years after surgery
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the 6-meter hop for time.
Knee Outcome Survey Activities of Daily Living (KOS-ADLS) Scale | At 2 years after surgery
  The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability. This scale would be appropriate for patients who either do not participate in sports or recreational activities or for those who have not yet progressed to performing these activities
Knee Outcome Survey Activities of Daily Living (KOS-ADLS) Scale | At 5 years after surgery
  The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability. This scale would be appropriate for patients who either do not participate in sports or recreational activities or for those who have not yet progressed to performing these activities
Knee Outcome Survey Activities of Daily Living (KOS-ADLS) Scale | At 10 years after surgery
  The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability. This scale would be appropriate for patients who either do not participate in sports or recreational activities or for those who have not yet progressed to performing these activities
Knee laxity | At 5 years after surgery
  The side to side knee joint laxity of patients after anterior cruciate ligament surgery can be divided into four grades: grade A: -1~2mm(0+), grade B: 3~5mm (1+), grade C: 6~10mm (2+) and D Grade: >10mm(3+) assessed by Lachman test of physical examination.
Knee laxity | At 10 years after surgery
  The side to side knee joint laxity of patients after anterior cruciate ligament surgery can be divided into four grades: grade A: -1~2mm(0+), grade B: 3~5mm (1+), grade C: 6~10mm (2+) and D Grade: >10mm(3+) assessed by Lachman test of physical examination.
Quadriceps strength | At 5 years after surgery
  Side to side quadriceps strength assessed by Biodex arthrometer test
Quadriceps strength | At 10 years after surgery
  Side to side quadriceps strength assessed by Biodex arthrometer test
Lysholm score | At 2 years after surgery
  Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 5 years after surgery
  Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 10 years after surgery
  Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 2 years after surgery
  Patients will be asked to fill out the KOOS score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 5 years after surgery
  Patients will be asked to fill out the KOOS score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 10 years after surgery
  Patients will be asked to fill out the KOOS score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 5 years after surgery
  Patients will be asked to fill out the IKDC2000 score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 10 years after surgery
  Patients will be asked to fill out the IKDC2000 score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Tegner Score | At 2 years after surgery
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Tegner Score | At 5 years after surgery
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Tegner Score | At 10 years after surgery
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Short Form (SF)-36,The medical outcome study 36-items short form health survey (SF-36) | At 2 years after surgery
  Patients will be asked to fill out the SF-36 to document the quality of life . General health-related quality of life: SF-36 physical component score (range 0 to 100; higher score = better health state) at 2 yearsTh minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Short Form (SF)-36 ,The medical outcome study 36-items short form health survey (SF-36) | At 5 years after surgery
  Patients will be asked to fill out the SF-36 to document the quality of life.General health-related quality of life: SF-36 physical component score (range 0 to 100; higher score = better health state) at 5 years. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Short Form (SF)-36,The medical outcome study 36-items short form health survey | At 10 years after surgery
  Patients will be asked to fill out the SF-36 to document the quality of life.General health-related quality of life: SF-36 physical component score (range 0 to 100; higher score = better health state) at 10 years. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Magnetic resonance imaging (MRI) | At 5 years after surgery
  The difference in signal density between reconstructed ACL and PCL was used to measure graft ligamentation on MRI. Higher signal values represent higher inflammation and lower signal values represent better ligamentation.
Magnetic resonance imaging (MRI) | At 10 years after surgery
  The difference in signal density between reconstructed ACL and PCL was used to measure graft ligamentation on MRI. Higher signal values represent higher inflammation and lower signal values represent better ligamentation.
Knee laxity （KT-2000 arthrometer） | At 5 years after surgery
  The knee laxity test of the forward KT-2000 measured knee laxity at pressures of 132Nt, 88Nt, 66Nt, and 44Nt, respectively, while the back-pushing KT-2000 was measured at -132NT, 88Nt, 66Nt, and -44Nt. The foward-pushing KT-2000 asessed side-to-side can be stratified into five levels are (A) < - 1 mm, (B) - 1 to 1 mm, (C) 1-3 mm, (D) 3-5 mm and (E) > 5 mm.
  The back-pushing KT-2000 is also divided into side to side differences as (A) < - 2 mm, (B) - 2 to - 0.5 mm, (C) - 0.5 to 0.5 mm, (D) 0.5-1 mm and ( E) > 1 mm.
Knee laxity （KT-2000 arthrometer） | At 10 years after surgery
  The knee laxity test of the forward KT-2000 measured knee laxity at pressures of 132Nt, 88Nt, 66Nt, and 44Nt, respectively, while the back-pushing KT-2000 was measured at -132NT, 88Nt, 66Nt, and -44Nt. The foward-pushing KT-2000 asessed side-to-side can be stratified into five levels are (A) < - 1 mm, (B) - 1 to 1 mm, (C) 1-3 mm, (D) 3-5 mm and (E) > 5 mm.
  The back-pushing KT-2000 is also divided into side to side differences as (A) < - 2 mm, (B) - 2 to - 0.5 mm, (C) - 0.5 to 0.5 mm, (D) 0.5-1 mm and ( E) > 1 mm.
Computed tomography (CT) | At 1 days after surgery.(baseline)
  Computed tomography was used to acquire a baseline of the bone tunnel one days after ACL reconstruction for comparison in studies of bone tunnel widening at follow-up visits.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Xu Z, Song S, Mao Z, Huang X, Luo M, Zhou X, Xu B, Ye J, Song Y, Yu J. Which technique provides more benefits in return to sports and clinical outcomes after anterior cruciate ligament reconstruction: Double-bundle or single-bundle? A randomized controlled study. Chin Med J (Engl). 2025 Sep 20;138(18):2283-2292. doi: 10.1097/CM9.0000000000003267. Epub 2024 Oct 10. PMID 39385323